CLINICAL TRIAL: NCT05627297
Title: Artificial Intelligence to Optimize Early-stage Hepatocellular CarcinomaTreatment Based on Multi-modal Image
Brief Title: Applying Artificial Intelligence to Optimize Early-stage Hepatocellular Carcinoma Treatment Based on Multi-modal Image
Acronym: AI-HCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: WentaoKong
Record Dates: First submitted 2022-11-16; First posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SR
  Interventions: Other: CEUS and CEMRI
- RFA
  Interventions: Other: CEUS and CEMRI

INTERVENTIONS:
Other: CEUS and CEMRI — contrast-enhanced ultrasound and contrast-enhanced MRI examination

SUMMARY:
This study intends to establish two prognostic models based on contrast-enhanced ultrasound (CEUS) and dynamic enhanced magnetic resonance (DE-MRI) multimodal images: prognostic model of liver cancer patients after hepatectomy and prognostic model of liver cancer patients after radiofrequency ablation. Combined with artificial intelligence imaging omics, traditional imaging omics and clinical information, to predict and compare the prognosis of two different treatment methods for early liver cancer, so as to realize the individual selection of treatment methods for early liver cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Primary single hepatocellular carcinoma confirmed by histology or cytology, with a maximum diameter ≤5.0 cm;

  * Good liver function, Child-Pugh grade A;

    * No serious dysfunction of heart, lung, kidney and other important organs ④ Liver resection or radiofrequency ablation was performed in our hospital, and the study protocol and follow-up procedure were followed.

Exclusion Criteria:

* Patients who cannot perform DCE-MRI examination due to metal implants in the body ② Patients who had received other treatment before DCE-MRI or CEUS;

  * Invisible lesions, diffuse lesions or poor DCE-MRI/CEUS image quality under CEUS; ④ Drug abuse, clinical or psychological or social factors that make informed consent or study implementation affected.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 200
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Good/Poor overall survival | 2022/12/01-2025/12/01

CONTACTS AND LOCATIONS:
Overall Officials: Wentao Kong, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No